CLINICAL TRIAL: NCT02228655
Title: An Exploratory, Uncontrolled, Open-labeled Trial to Evaluate the Effect of FMX-8 Treatment for Anemia in Patients With Chronic Kidney Disease (CKD), Stage 4 or 5
Brief Title: An Exploratory Study to Evaluate FMX-8 to Treat Anemia in CKD
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Inability to recruit patients meeting eligibilty criteria.
Sponsor: FerruMax Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX-C-888
Record Dates: First submitted 2014-07-17; First posted 2014-08-29 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Anemia in Chronic Kidney Disease
Keywords: Chronic Kidney Disease; CKD; Anemia of Chronic Illness
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FMX-8 (Other): FMX-8 for injection, 15mg/kg, twice weekly, 29 days
  Interventions: Drug: FMX-8

INTERVENTIONS:
Drug: FMX-8

SUMMARY:
FMX-8 is a new type of drug being tested for the treatment of anemia in chronic illnesses.

ELIGIBILITY:
Inclusion Criteria:

* a documented hemoglobin level to be less than 10 g/dL at screening
* diagnoses of CKD 4 or 5
* body mass index (BMI) between 18 kg/m2 and 42 kg/m2, inclusive, based upon the height and weight at screening
* ferritin levels ≥100 ng/ml or Tsat ≥20% at screening
* erythropoietin (EPO) level greater than 8 ng/mL
* able to provide written informed consent
* able to understand and follow all trial procedures
* willing to use contraception as detailed in the protocol

Exclusion Criteria:

* receipt of red blood cell (RBC) transfusion within four weeks before screening
* overt gastrointestinal bleeding or other bleeding episode that required transfusion within 2 months prior to screening
* infection necessitating antibiotic or anti-viral treatment within a month prior to screening
* requiring Coumadin (warfarin), Pradaxa®, Eliquis®, or Xarelto®
* hemoglobinopathies such as homozygous sickle-cell disease or thalassemias of all types
* active hemolysis or chronic hypoxia
* active malignant diseases (except non-melanoma skin cancer) or life expectancy less than 6 months
* chronic, uncontrolled or symptomatic inflammatory disease or non-renal cause of anemia such as rheumatoid arthritis, systemic lupus erythematosus, HIV, or systemic acute infection
* on immunosuppressive therapeutics except topical corticosteroids or nasal sprays
* chronic congestive heart failure (New York Heart Association Class III, IV)
* significant hypertension (≥90 diastolic) based on a sitting diastolic blood pressure at screening
* kidney transplant within the past year: patients who are off immunosuppressive agents following a failed transplant are eligible for the trial
* end-stage liver disease
* known hypersensitivity to recombinant protein therapies
* female patients who are pregnant or breast feeding
* previous exposure to FMX-8
* previous exposure to Epogen®, Procrit® (erythropoietin) Aranesp® (darbepoietin alpha), Omontys® or Hematide® (peginesatide) anemia treatment
* uncontrolled hyperparathyroidism (PTH >750) based upon latest PTH determination within the past 4 months
* inability to comply with the trial scheduled visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin concentration | 57 day evaluation period

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Lecker, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Babitt JL, Huang FW, Wrighting DM, Xia Y, Sidis Y, Samad TA, Campagna JA, Chung RT, Schneyer AL, Woolf CJ, Andrews NC, Lin HY. Bone morphogenetic protein signaling by hemojuvelin regulates hepcidin expression. Nat Genet. 2006 May;38(5):531-9. doi: 10.1038/ng1777. Epub 2006 Apr 9. PMID 16604073
- [Background] Babitt JL, Huang FW, Xia Y, Sidis Y, Andrews NC, Lin HY. Modulation of bone morphogenetic protein signaling in vivo regulates systemic iron balance. J Clin Invest. 2007 Jul;117(7):1933-9. doi: 10.1172/JCI31342. PMID 17607365
- [Background] Huang FW, Pinkus JL, Pinkus GS, Fleming MD, Andrews NC. A mouse model of juvenile hemochromatosis. J Clin Invest. 2005 Aug;115(8):2187-91. doi: 10.1172/JCI25049. PMID 16075059
- [Background] KDOQI. KDOQI Clinical Practice Guideline and Clinical Practice Recommendations for anemia in chronic kidney disease: 2007 update of hemoglobin target. Am J Kidney Dis. 2007 Sep;50(3):471-530. doi: 10.1053/j.ajkd.2007.06.008. No abstract available. PMID 17720528
- [Background] Theurl I, Schroll A, Sonnweber T, Nairz M, Theurl M, Willenbacher W, Eller K, Wolf D, Seifert M, Sun CC, Babitt JL, Hong CC, Menhall T, Gearing P, Lin HY, Weiss G. Pharmacologic inhibition of hepcidin expression reverses anemia of chronic inflammation in rats. Blood. 2011 Nov 3;118(18):4977-84. doi: 10.1182/blood-2011-03-345066. Epub 2011 Jul 5. PMID 21730356
- [Background] Weiss G, Goodnough LT. Anemia of chronic disease. N Engl J Med. 2005 Mar 10;352(10):1011-23. doi: 10.1056/NEJMra041809. No abstract available. PMID 15758012
- [Background] Weiner DE. Causes and consequences of chronic kidney disease: implications for managed health care. J Manag Care Pharm. 2007 Apr;13(3 Suppl):S1-9. doi: 10.18553/jmcp.2007.13.s3.1. PMID 17402808